CLINICAL TRIAL: NCT02483793
Title: Randomized Prospective Trial Comparing Oxybutynin and Tamsulosin for Stent Discomfort in the Pediatric Population
Brief Title: Prospective Trial Comparing Oxybutynin and Tamsulosin for Stent Pain in the Pediatric Population
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was withdrawn prior to IRB approval and prior to enrollment. The study was never opened, and no participants were enrolled.
Sponsor: Phoenix Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 15-065
Record Dates: First submitted 2015-06-22; First posted 2015-06-29 (Estimated); Last update posted 2026-01-14 (Actual); Status verified 2015-06

CONDITIONS: Disorder of Urinary Stent
MeSH Terms: interventions — Tamsulosin; oxybutynin

ARMS (2):
- Oxybutynin group (Active Comparator): This group will be prescribed oxybutynin as well as standard narcotic pain medications. Oxybutynin will be prescribed based off of standard dosing. Patients who are unable to swallow pills will be given oxybutynin elixir (0.5mg/kg/day, divided TID). Patients who are able to swallow pills will be given oxybutynin 5mg either BID or TID.
  Interventions: Drug: Oxybutynin
- Tamsulosin group (Active Comparator): This group will be prescribed tamsulosin and standard narcotic pain medication. Patients will be given tamsulosin 0.4mg at bedtime. This dosage has been used in other studies for children age ≥ 4.
  Interventions: Drug: Tamsulosin

INTERVENTIONS:
Drug: Tamsulosin
  Arms: Tamsulosin group
Drug: Oxybutynin
  Arms: Oxybutynin group

SUMMARY:
The primary objective of this study is to evaluate the efficacy and safety tamsulosin in reducing stent discomfort in the pediatric population in the peri-operative period. The secondary objective is to compare the efficacy of tamsulosin with that of oxybutynin in reducing stent discomfort.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 4-18 years will be enrolled in this study. We will include all patients who will have a ureteral stent placement after their procedure.

Exclusion Criteria:

* Patients with developmental delay or unable to verbalize their pain level will be excluded.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2015-07; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Number of doses of pain in medication used | 5 days post-op
  After surgery, each child will be prescribed the standard dosage of oxycodone/acetaminophen based on their weight. We will have the patient's family record the number of doses of narcotics used from post-operative day #1 to post-operative day #5 to assess their pain needs.
Pain scale based on the faces pain score | 5 days post-op
  We will have the family members record the child's pain score in the morning and evening using the faces pain scale and record the score.